CLINICAL TRIAL: NCT02057380
Title: A Phase II Open-label Rollover Study for Subjects That Have Participated in an Astellas Sponsored Linsitinib Trial
Brief Title: A Rollover Study for Subjects That Have Participated in an Astellas Sponsored Linsitinib Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7487-CL-0209; 2013-004076-34 (EudraCT Number)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumors
Keywords: Paclitaxel; Linsitinib; OSI-774; Advanced Solid Tumor; Tarceva; Erlotinib; OSI-906
MeSH Terms: interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol; Erlotinib Hydrochloride; Paclitaxel; Bortezomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- Arm A: High dose linsitinib twice daily monotherapy (Experimental): Arm A includes subjects from Protocol OSI-906-301
  Interventions: Drug: linsitinib
- Arm B: High dose linsitinib BID plus high dose erlotinib QD (Experimental): Arm B includes subjects from Protocol OSI-906-205
  Interventions: Drug: linsitinib; Drug: erlotinib
- Arm C: High dose erlotinib monotherapy once daily (Experimental): Arm C includes subjects from Protocol OSI-906-205 and OSI-906-207
  Interventions: Drug: erlotinib
- Arm D: High dose linsitinib BID plus weekly paclitaxel (Experimental): Arm D includes subjects from Protocol OSI-906-202
  Interventions: Drug: linsitinib; Drug: paclitaxel
- Arm E: Highest dose linsitinib intermittent once daily (Experimental): Arm E includes subjects from Protocol OSI-906-202, linsitinib on Days 1-3 of each week plus weekly paclitaxel
  Interventions: Drug: linsitinib; Drug: paclitaxel
- Arm F: Paclitaxel alone weekly (Experimental): Arm F includes subjects from Protocol OSI-906-202
  Interventions: Drug: paclitaxel
- Arm G: Lowest dose linsitinib twice daily + low dose erlotinib (Experimental): Arm G includes subjects from Protocol OSI-906-103
  Interventions: Drug: linsitinib; Drug: erlotinib
- Arm H: high dose linsitinib twice daily (Experimental): includes subjects from protocols SARC 022/CTEP 8945, linsitinib x28 days (each cycle)
  Interventions: Drug: linsitinib
- Arm I: highest dose linsitinib once daily (Experimental): includes subjects from EuroSARC protocol, linsitinib on Days 1-3; Days 8-10 and Days 15-17
  Interventions: Drug: linsitinib
- Arm J: Low dose linsitinib 2x daily+bortezomib & dexamethasone (Experimental): includes subjects from protocol MM-001; Days 1, 4, 8 & 11 (cycles 1-8) and Days 1, 8, 15 & 22 (cycles 9+)
  Interventions: Drug: linsitinib; Drug: Bortezomib; Drug: Dexamethasone
- Arm K: med. dose linsitinib 2x daily+bortezomib&dexamethasone (Experimental): includes subjects from protocol MM-001; Days 1, 4, 8 & 11 (cycles 1-8) and Days 1, 8, 15 & 22 (cycles 9+)
  Interventions: Drug: linsitinib; Drug: Bortezomib; Drug: Dexamethasone
- Arm L: high dose linsitinib 2x daily+bortezomib&dexamethasone (Experimental): includes subjects from protocol MM-001; Days 1, 4, 8 & 11 (cycles 1-8) and Days 1, 8, 15 & 22 (cycles 9+)
  Interventions: Drug: linsitinib; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: linsitinib — oral
  Other Names: OSI-906
  Arms: Arm A: High dose linsitinib twice daily monotherapy; Arm B: High dose linsitinib BID plus high dose erlotinib QD; Arm D: High dose linsitinib BID plus weekly paclitaxel; Arm E: Highest dose linsitinib intermittent once daily; Arm G: Lowest dose linsitinib twice daily + low dose erlotinib; Arm H: high dose linsitinib twice daily; Arm I: highest dose linsitinib once daily; Arm J: Low dose linsitinib 2x daily+bortezomib & dexamethasone; Arm K: med. dose linsitinib 2x daily+bortezomib&dexamethasone; Arm L: high dose linsitinib 2x daily+bortezomib&dexamethasone
Drug: erlotinib — oral
  Other Names: OSI-774; Tarceva
  Arms: Arm B: High dose linsitinib BID plus high dose erlotinib QD; Arm C: High dose erlotinib monotherapy once daily; Arm G: Lowest dose linsitinib twice daily + low dose erlotinib
Drug: paclitaxel — Intravenous (IV) infusion
  Arms: Arm D: High dose linsitinib BID plus weekly paclitaxel; Arm E: Highest dose linsitinib intermittent once daily; Arm F: Paclitaxel alone weekly
Drug: Bortezomib — Subcutaneous or IV
  Other Names: Velcade
  Arms: Arm J: Low dose linsitinib 2x daily+bortezomib & dexamethasone; Arm K: med. dose linsitinib 2x daily+bortezomib&dexamethasone; Arm L: high dose linsitinib 2x daily+bortezomib&dexamethasone
Drug: Dexamethasone — IV, Oral
  Other Names: Maxidex; Baycadron; Ozurdex; Decadron
  Arms: Arm J: Low dose linsitinib 2x daily+bortezomib & dexamethasone; Arm K: med. dose linsitinib 2x daily+bortezomib&dexamethasone; Arm L: high dose linsitinib 2x daily+bortezomib&dexamethasone

SUMMARY:
The purpose of this study is to provide access to continued treatment for subjects who participated in other Astellas sponsored trials and for whom the investigator feels the subject may benefit from continued treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject must currently be participating in an Astellas sponsored linsitinib trial that has ended with respect to the overall study analysis.
* Subject must not have met criteria for discontinuation or have progressed on the current linsitinib study in which they are participating.
* Subject must be deriving benefit from continued treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04-16 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (12):
- United States (5):
  - Site US10004, La Jolla, California
  - Site US10006, Tampa, Florida
  - Site US10002, Baltimore, Maryland
  - Site US10008, Ann Arbor, Michigan
  - Site US10001, Oklahoma City, Oklahoma
- Site BR55005, Porto Alegre, Rio Grande do Sul, Brazil
- Site CZ42001, Ostrava-Poruba, Czechia
- Germany (2):
  - Site DE49002, Berlin
  - Site DE49001, Würzburg
- Site PL48001, Szczecin, West Pomeranian Voivodeship, Poland
- Site SG65002, Singapore, Singapore
- Site TH66003, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=252